CLINICAL TRIAL: NCT01994785
Title: Does the Use of Capnography in Routine EGD and Colonoscopy Targeting Moderate Sedation With a Benzodiazepine and Opioid Improve Safety?
Brief Title: Use of Capnography in EGD and Colonoscopy With Moderate Sedation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, John Vargo, Department Chairman, Gastroenterology and Hepatology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CC-13-792
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Hypoxia; Apnea; Hypotension; Hypopnea
Keywords: Sedation; Endoscopy; Capnography
MeSH Terms: conditions — Hypoxia; Apnea; Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EGD capnography open (Active Comparator): Capnographic monitoring during EGD - Data made available to study staff throughout procedure
  Interventions: Diagnostic Test: Capnographic Monitoring
- EGD capnography blinded (Active Comparator): Capnographic monitoring during EGD - Data made available to study staff only if necessary for safety reasons
  Interventions: Diagnostic Test: Capnographic Monitoring
- Colonoscopy capnography open (Active Comparator): Capnographic monitoring during Colonoscopy - Data made available to study staff throughout procedure
  Interventions: Diagnostic Test: Capnographic Monitoring
- Colonoscopy capnography blinded (Active Comparator): Capnographic monitoring during Colonoscopy - Data made available to study staff only if necessary for safety reasons
  Interventions: Diagnostic Test: Capnographic Monitoring

INTERVENTIONS:
Diagnostic Test: Capnographic Monitoring — Capnographic Monitoring: Patients will undergo procedures with real-time capnographic monitoring

SUMMARY:
This study will provide capnography monitoring during routine upper endoscopy and colonoscopy with moderate sedation in order to see if it improves safety.

DETAILED DESCRIPTION:
The majority of gastrointestinal endoscopic procedures currently performed in the United States are done under moderate sedation, primarily utilizing the combination of an opioid and benzodiazepine. The endoscopy team administers the medications, most commonly the endoscopy nursing team at the discretion of the endoscopist, with careful cardiopulmonary monitoring during the procedure. The use of sedation can lead to serious unplanned adverse events. Cardiopulmonary events related to the use of sedation in GI endoscopy include hypotension, hypoxia, and hypopnea/apnea. The most common of these adverse events is hypoxia, which can occur in 10-70% of patients. Although most of these events are transient and respond to supplemental oxygenation, studies have shown electrocardiographic signs of cardiac ischemia in patients with no known preexisting heart disease. Pulse oximetry can help detect hypoxia related to perfusion deficits (cardiac) or ventilation factors (respiratory) however, it is not designed to detect ventilator precursors of alveolar hypoventilation, which primarily present as decreased respiratory rate or hypopnea/apnea.

Capnography utilizes the near-infrared spectrophotometric absorption spectrum of carbon dioxide (CO2) at 420 nm to provide graphic assessment of the ventilation status via the partial pressure of carbon dioxide during the respiratory cycle. Previous studies have shown it to improve safety by detecting early indicators of hypoxia and/or signs of alveolar hypoventilation. Studies have shown that when targeting deep sedation in advanced endoscopic procedures utilizing capnography was superior to pulse oximetry alone in detecting respiratory depression. There is also evidence that shows utilizing capnography in advanced endoscopic procedures significantly decreased the incidence of hypoxia versus standard monitoring with the procedural team blinded to the capnographic data (132 blinded vs. 49 open, P<.001) and rates of hypoxia (69% blinded vs. 46% open, P<.001) were significantly lower with capnography monitoring.

Routine esophagogastroduodenoscopy (EGD) and colonoscopy with moderate sedation is safe with rates of sedation associated adverse events occurring in 8 per 100,000 cases. Lightdale and colleagues showed in a prospective, double blinded randomized controlled trial in a pediatric population undergoing routine EGD or colonoscopy targeting moderate sedation with opioid-benzodiazepine combinations that patients in the intervention capnography arm were less likely (4% vs. 20%, P<.03) to have an intra-procedural episodes of hypoxia (defined as SpO2<95% for >5sec). No adverse events related to episodes of hypoxia were reported in this trial, but it was underpowered to evaluate this outcome. To our knowledge, there is no data on use of capnography in adult patients undergoing EGD and colonoscopy targeting moderate sedation with the combination of an opioid and benzodiazepine.

The American Society of Anesthesiology (ASA) has recently updated their standards for basic anesthetic monitoring to now state that during moderate sedation all patients should have capnographic monitoring. This was updated from the previous standards for basic monitoring that stated capnography could be used during these levels of sedation. This is a significant change in the practice model for monitoring patients undergoing routine endoscopy with moderate sedation and, as the standards for basic monitoring are often used as a basis for regulatory guidelines applied to hospital or ambulatory care centers, the addition of requiring capnographic monitoring changes the landscape of procedural sedation for gastrointestinal endoscopy across the United States. The evidence cited for this update in monitoring guidelines included the Lightdale pediatric endoscopy study and our groups study that utilized capnography in advanced endoscopic procedures. There was no data available in adult patients undergoing routine EGD or colonoscopy at the time of the updated guidelines. The extrapolation of advanced endoscopic procedures to routine endoscopy is of limited use as the procedures are targeting different levels of sedation (deep vs. moderate, respectively) and the length of the procedures is significantly different.

The rationale for not using capnography in moderate sedation arises from its ability to lead to false alarms, such as pseudo-apnea secondary to swallowing or failure to monitor both the oral and nasal airways for respiratory activity, as some patients will transition to nasal or mouth breathing during sedation. These alarms during a procedure may lead to interruption, delay, or early termination. Increased costs for capnography equipment and having appropriately trained endoscopy team members to interpret capnography results will be difficult to accomplish with no patient data supporting the effectiveness of its use in routine EGD and colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* >18yrs with full decision making capacity
* Scheduled for elective upper endoscopy or colonoscopy with moderate sedation

Exclusion Criteria:

* ASAPS class III or higher.
* History of a demonstrated allergy or intolerance to a benzodiazepine or opioid
* Patients scheduled for both upper endoscopy and colonoscopy during the same endoscopy day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Vargo, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Independence, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta PP, Kochhar G, Albeldawi M, Kirsh B, Rizk M, Putka B, John B, Wang Y, Breslaw N, Lopez R, Vargo JJ. Capnographic Monitoring in Routine EGD and Colonoscopy With Moderate Sedation: A Prospective, Randomized, Controlled Trial. Am J Gastroenterol. 2016 Mar;111(3):395-404. doi: 10.1038/ajg.2015.437. Epub 2016 Feb 23. PMID 26902229

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EGD Capnography Open | EGD Capnography Blinded | Colonoscopy Capnography Open | Colonoscopy Capnography Blinded
Started | 109 | 109 | 117 | 117
Completed | 101 | 108 | 117 | 114
Not Completed | 8 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EGD Capnography Open | EGD Capnography Blinded | Colonoscopy Capnography Open | Colonoscopy Capnography Blinded | Total
Number analyzed (Participants) | 101 | 108 | 117 | 114 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (17.3) | 49.8 (17.0) | 54.1 (13.8) | 55.3 (13.3) | 54.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 58 | 59 | 251
  Male | 36 | 39 | 59 | 55 | 189
Region of Enrollment [Number; unit: participants]
  United States | 101 | 108 | 117 | 114 | 440

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Hypoxia During Capnography Monitoring.
Time Frame: One day--data is collected during one endoscopic procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | EGD Capnography Open | EGD Capnography Blinded | Colonoscopy Capnography Open | Colonoscopy Capnography Blinded
Number analyzed (Participants) | 109 | 109 | 117 | 117
Participants | 54 | 59 | 61 | 63

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of initial sedation until participants were cleared to return home following their study endoscopic procedure
Arm/Group | EGD Capnography Open | EGD Capnography Blinded | Colonoscopy Capnography Open | Colonoscopy Capnography Blinded
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/108 | 0/117 | 0/114
Other Adverse Events (participants affected / at risk) | 0/101 | 0/108 | 0/117 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes